CLINICAL TRIAL: NCT04035057
Title: Examining Behavioral Strategies for Enhancing Therapists' Delivery of Exposure Therapy
Acronym: STRIVE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bradley Hospital (Other)
Responsible Party: Principal Investigator, Joshua Kemp, Principal Investigator, Bradley Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: R34MH118199 (NIH)
Record Dates: First submitted 2019-04-29; First posted 2019-07-29 (Actual); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Anxiety Disorders
Keywords: Therapist Training; Exposure Therapy; Experimental Therapeutics
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Two phases: Phase I is a case-series analysis to determine the necessary dosage to engage the training intervention target (i.e., therapist negative beliefs). Phase II is a randomized trial of a behaviorally-enhanced training versus standard didactic training.
Who Masked: Participant
Masking Description: Therapist participants who are completing the training intervention are blind to the other training condition
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behaviorally Enhanced Training Strategies (Experimental): Both training conditions will receive a 1.5 day training followed by ongoing supervision while they implement exposure therapy with patients recruited to the study. The first full day will consist of the same foundational information in both conditions. The two conditions will differ in their training focus during the subsequent half-day training. The Behaviorally Enhanced condition will involve therapist engagement in repeated self-exposure and partner-exposure exercises with the goal of targeting and reducing therapists' reservations about using exposure with their patients. The focus of ongoing supervision following the initial 1.5 day training workshop will also differ by condition. The Behaviorally Enhanced condition will include regular sampling and feedback on therapists' remaining reservations about exposure in additional to counseling the implementation of exposure with therapists' patients.
  Interventions: Other: Behaviorally Enhanced Training
- Standard Didactic Training (Active Comparator): Both training conditions will receive a 1.5 day training followed by ongoing supervision while they implement exposure therapy with patients recruited to the study. The first full day will consist of the same foundational information in both conditions.The two conditions will differ in their training focus during the subsequent half-day training. The Standard Didactic condition will involve additional didactic instruction related to common barriers and more advanced delivery concepts than will be presented in the half-day training for the Behaviorally Enhanced condition. The focus of ongoing supervision following the initial 1.5 day training workshop will also differ by condition. The Standard Didactic condition will involve counseling on the implementation of exposure with therapists' patients without explicit focus on therapists' remaining reservations about exposure.
  Interventions: Other: Standard Didactic Training

INTERVENTIONS:
Other: Behaviorally Enhanced Training — Therapists in the Behaviorally Enhanced Training will receive the same didactic instruction as those in the Standard Didactic Training arm during the first full day of training. In the second half-day training, those in the Behaviorally Enhanced Training arm will focus on behavioral strategies (i.e., exposure to exposure) that provide direct experience with the process of treatment delivery.
  Arms: Behaviorally Enhanced Training Strategies
Other: Standard Didactic Training — Therapists in the Standard Didactic Training arm will complete training as usual, consisting of PowerPoint and video training tasks instructing the delivery of exposure therapy for anxious youth.
  Arms: Standard Didactic Training

SUMMARY:
The goal of this study is to test a targeted training for overcoming known barriers to the uptake and quality delivery of exposure therapy among community mental health providers. The first phase (Year 1) of the study is a case-series analysis of six therapists with the goal of determining whether the targeted training strategies (i.e., exposure to exposure) are capable of engaging therapists' reservations about exposure. Information from the first phase will be used to optimize the behavioral training strategies to be tested in the second phase. The second phase (Years 2 & 3) will be a randomized trial of training conditions comparing Behaviorally Enhanced Training Strategies to a Standard Didactic Training. After an initial workshop training, therapists in the second phase will receive ongoing consultation while they deliver exposure therapy with their anxious patients. Sessions will be video-recorded and therapist behaviors will be coded to assess for differences in the manner in which exposure is delivered between training conditions.

DETAILED DESCRIPTION:
Following decades of psychosocial treatment research the field has established numerous evidence-based practices (EBPs) for mental disorders, but has struggled to widely disseminate these practices in community settings. Exposure therapy for anxiety disorders represents one of the most glaring examples of this research to practice gap. A well-known barrier to the dissemination and quality delivery of exposure therapy is therapists' negative beliefs about its potential danger or intolerability for patients. These beliefs are common even among therapists who report receiving specialized training; thus, research is needed to develop targeted training strategies for reducing negative beliefs and improving delivery quality. Preliminary research suggests specific behavioral strategies (i.e., self-exposure) may reduce negative beliefs above and beyond standard didactic trainings (Farrell, Kemp et al., 2016). Building upon these findings, the investigators propose a novel experimental therapeutics approach to developing and testing a targeted behavioral training for augmenting negative beliefs in a sample of community mental health professionals. The first phase of the study is a case-series analysis for establishing target engagement (i.e., belief reduction) and determining adequate dosing of the behavioral strategies. Phase two is a randomized trial of the behaviorally-enhanced training strategies (BeTS) against a standard didactic protocol. Therapist will complete a day-long workshop followed by weekly consultation while delivering exposure for children with anxiety disorders. In-session delivery behavior will be recorded and examined using a validated micro-analytic coding system. It is hypothesized that therapists in the BeTS condition will evidence significantly lower negative beliefs about exposure relative to the didactic condition, at 1) post-workshop, and 2) end of study. IT is also hypothesized that the degree of negative belief reduction following the initial workshop training will be associated with 1) higher rates of optimal in-session delivery behaviors, and 2) lower rates of suboptimal delivery behaviors as measured by both self-report and observational coding data. This study will establish an innovative model for developing a targeted training intervention capable of increasing the dissemination and quality of exposure therapy and other EBPs.

ELIGIBILITY:
Inclusion Criteria: Therapists

* Agency hours >8 hours a week.

Exclusion Criteria:

* Training procedure are unacceptable to therapist

Patient Participants: Age 5 - 17 years

Inclusion Criteria:

* Primary or co-primary diagnosis of Separation Anxiety Disorder, Specific Phobia, Social Anxiety Disorder, Panic Disorder, or OCD
* Children < age 12 have a caretaker available to participate in treatment
* Patient and at least one parent are English speaking

Exclusion Criteria:

* Concurrent psychotherapy for treatment of anxiety
* Psychosis, Pervasive Developmental Disorder, or Mental Retardation.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in therapist reservations about exposure | Baseline (pre-workshop) & End of the 1.5 day Training Workshop
  The Therapist Beliefs about Exposure (TBES) will be administered to assess the extent to which therapists harbor negative perceptions of exposure therapy and its tolerability among their patients. The TBES is a 21-item scale with a 0 ("Disagree Strongly") to 4 ("Strongly Agree") rating scale. TBES scores are summed and range from 0 to 84, with lower scores indicating less reservations.
Change in therapist reservations about exposure | End of 1.5 day Training Workshop & End of Therapist Participation in the Study, on average 1 year.
  The Therapist Beliefs about Exposure (TBES) will be administered to assess the extent to which therapists harbor negative perceptions of exposure therapy and its tolerability among their patients. The TBES is a 21-item scale with a 0 ("Disagree Strongly") to 4 ("Strongly Agree") rating scale. TBES scores are summed and range from 0 to 84, with lower scores indicating less reservations.
Therapist Delivery Behavior | The first 12 exposure sessions with patients recruited to the study will be videotaped and coded, on average 3 months.
  We will apply a validated microanalytic coding system to determine the extent to which therapists' in-session behavior aligns with indicators of "optimal" and "suboptimal" delivery. Videotaped delivery behaviors are coded and time-stamped. Categories of delivery behavior are then summed within and across sessions.

SECONDARY OUTCOMES:
Change in Patients' Symptoms of Anxiety | Independent raters will administer the PARS at pre-treatment and post-treatment, on average 3 months
  Patients with symptoms of anxiety will be administered the Pediatric Anxiety Rating Scale (PARS), which is a clinician-rated measure of anxiety symptom severity for use with multiple anxiety disorders. The measure consists of a symptom checklist and seven symptom severity items. The symptom severity items are rated using a 0 to 5 scale with lower ratings indicating less severity. Scores are summed and range from 0 to 35.
Change in Patients' Symptoms of Obsessive-Compulsive Disorder (OCD) | Independent raters will administer the CY-BOCS at pre-treatment and post-treatment, on average 3 months.
  Patients presenting with symptoms of OCD will be administered the Child Yale-Brown Obsessive-Compulsive Scales (CY-BOCS)61: the clinician-administered, "gold standard" assessment of OCD symptom severity with excellent psychometric properties. Total scores for obsession and compulsion subscales range from 0 (no symptoms) to 40 (severe).

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Kemp, PhD, Principal Investigator — Bradley Hospital
Locations (1):
- Bradley Hospital, Riverside, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures, but not raw coding data, will be made available.
Supporting Information: Study Protocol
Time Frame: Data will be available within 6 months of study completion.
Access Criteria: Data access requests will be reviewed by an external Independent Review Panel. Requestors will be required to sign a Data Access Agreement.